CLINICAL TRIAL: NCT01364467
Title: The Effect of Oral Guaifenesin on Pediatric Chronic Rhinitis: A Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM13538
Record Dates: First submitted 2011-05-04; First posted 2011-06-02 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Chronic Rhinitis
MeSH Terms: interventions — Guaifenesin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo is provided by the sponsor and is identical in composition to the treatment only lacking active drug.
  Interventions: Drug: Placebo
- Guaifenesin (Active Comparator)
  Interventions: Drug: Guaifenesin

INTERVENTIONS:
Drug: Placebo — Children aged 7-11 years old will receive placebo 200 mg three times a day (TID), while children older than 12 will receive Placebo 400 mg TID.
  Arms: Placebo
Drug: Guaifenesin — Children aged 7-11 years old will receive guaifenesin 200 mg TID, while children older than 12 will receive guaifenesin 400 mg TID.
  Arms: Guaifenesin

SUMMARY:
This is a 14-day, randomized, placebo-controlled, parallel group, masked clinical trial of oral guaifenesin for the therapy of Chronic Rhinitis (CRS) in 36 children between the ages of 7 and 18 years. The study investigates the effectiveness of guaifenesin in the relief of nasal symptoms in children with CRS using the sinonasal 5 survey (SN-5) in comparison to nasal airway volume, and biophysical properties of nasal secretion. The investigators hypothesize that Guaifenesin use over a period of 14 days improves subjective nasal complaints in pediatric patients with chronic rhinitis and nasal congestion, as measured by the SN-5 survey compared to use of placebo. There will be an observed improvement in nasal volume and cross-sectional area following use of guaifenesin, and nasal secretions will have more favorable mucociliary and sneeze clearability compared to use of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 7 and 18 years, diagnosed with Chronic Rhinitis and nasal stuffiness for at least 3 month duration.

Exclusion Criteria:

* Children with immunodeficiency, cystic fibrosis, acute or subacute symptoms, signs of bacterial infection, and/or those who are unable to cooperate with testing will be excluded. Children with documented use of the study medication in the month before evaluation and during period of symptoms will also be excluded.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelley Dodson, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University Children's Hospital of Richmond, Children's Pavilion & Nelson Clinic, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Guaifenesin
Started | 10 | 20
Completed | 9 | 18
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Guaifenesin | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.75 (2.99) | 10.35 (2.9) | 10.46 (2.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 5 | 11 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 11 | 15
  White | 2 | 6 | 8
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 20 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in Subjective Nasal Scoring
Description: The Sinus and Nasal Quality of Life Survey (SN-5) questionnaire assesses the impact of infection on nasal symptoms, emotion, and activity. The SN-5 is a 5-item scale with each item rated on a scale of worsening symptoms from 1 (none of the time) through 7 (all of the time). Items were averaged to yield a single score ranging from 1 (better outcomes) to 7 (worse outcomes). Scores were used to asses change in disease severity and the impact of interventions on subjective complaints from baseline to follow-up.
Time Frame: Baseline to 10 Minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Guaifenesin
Number analyzed (Participants) | 9 | 18
score on a scale | 0.62 (0.59) | 1.53 (1.04)
Statistical Analysis 1: Comparison: Placebo vs Guaifenesin; Test type: Other; p = 0.013, t-test, 2 sided

2. Secondary Outcome: Nasal Volume
Description: Acoustic rhinometry is used to measure cross-sectional volume of the nasal cavity allowing the calculation of nasal volume.
Time Frame: 15 Minutes
Measure: Mean (Standard Deviation); unit: Square centimeters
Arm/Group | Placebo | Guaifenesin
Number analyzed (Participants) | 9 | 18
Square centimeters
  Right nostril | 1.10 (0.4) | 1.13 (0.66)
  Left nostril | 0.83 (0.44) | 1.08 (0.67)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.98, t-test, 2 sided
Statistical Analysis 2: Comparison: Guaifenesin; Test type: Superiority; p = 0.65, t-test, 2 sided

3. Secondary Outcome: Nasal Secretion Collection
Description: To measure the biophysical properties of nasal secretions for improved mucus clearance.
Time Frame: 10 minutes
Population: Unable to analyze due to insufficient sample material
Arm/Group | Placebo | Guaifenesin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Placebo | Guaifenesin
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/18
Other Adverse Events (participants affected / at risk) | 0/9 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT01364467/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT01364467/SAP_001.pdf